CLINICAL TRIAL: NCT04511481
Title: Deep Learning Magnetic Resonance Imaging Radiomic Predict Platinum-sensitive in Patients With Epithelial Ovarian Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Herui Yao, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2020-072
Record Dates: First submitted 2020-08-11; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Predictive Cancer Model

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- platinum-resistant group
  Interventions: Other: Radiomic Algorithm
- platinum-sensitive group
  Interventions: Other: Radiomic Algorithm

INTERVENTIONS:
Other: Radiomic Algorithm — Different radiomic and machine learning strategies for radiomic features extraction, sorting features and model constriction

SUMMARY:
Platinum-sensitive is an important basis for the treatment of recurrent epithelial ovarian cancer (EOC) without effective methods to predict.We aimed to develop and validate the EOC deep learning system to predict the platinum-sensitive of EOC patients through analysis of enhanced magnetic resonance imaging (MRI) images before initial treatment.Ninety-three EOC patients received platinum-based chemotherapy (>= 4 cycles) and debulking surgery from Sun Yat-sen Memorial Hospitalin China from January 2011 to January 2020 were enrolled. This deep-learning EOC signature achieved a high predictive power for platinum-sensitive, and the signature based on MRI whole volume is better than that on primary tumor area only.

ELIGIBILITY:
Inclusion Criteria:

* (1)Patients with epithelial ovarian cancer (2 )Patients received platinum-based chemotherapy (>= 4 cycles) and debulking surgery

Exclusion Criteria:

* Patients with epithelial ovarian cancer received less than 4 cycles platinum-based chemotherapy or no debulking surgery

Ages: 22 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients received platinum-based chemotherapy (>= 4 cycles) and debulking surgery from Sun Yat-sen Memorial Hospital in China from January 2011 to January 2020
Sampling Method: Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-08-03 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Platinum sensitivity | 9 years
  Platinum sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The datasets used or analysed during the current study are available from the corresponding author on reasonable request.